CLINICAL TRIAL: NCT06769087
Title: Comparative Analysis of Clinical and Patient-Reported Outcomes: Immediate Versus Postoperative Day 1 Removal of Urinary Catheter After Colorectal Cancer Surgery in a Non-inferiority, Randomized Controlled Trial.
Brief Title: Comparing Immediate Removal and Postoperative 1 Day of Urinary Catheter After Colorectal Cancer Surgery
Acronym: POUR
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Eunpyeong St. Mary's Hospital, The Catholic University of Korea (Unknown); Catholic University of Korea, Yeouido St. Mary's Hospital (Unknown); The Catholic University of Korea Uijeongbu St.Marys Hostpial (Unknown); Saint Vincent's Hospital, Korea (Other); Incheon St.Mary's Hospital/The Catholic University (Unknown)
Responsible Party: Principal Investigator, Yoon Suk Lee, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KC24EISI0519; Seoul St.Mary's hospital (Other: Seoul St.Mary's hospital)
Record Dates: First submitted 2024-12-30; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer; Postoperative Complication; Urinary Retention Postoperative; Enhanced Recovery After Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: prospective, randomized controlled, non-inferior, multi-center trial
Who Masked: Participant, Investigator
Masking Description: Patients, care provider and surgeons will be unaware of randomized assignment until the end of surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate UC removal after surgery (Experimental): A urinary catheter is removed immediately after surgery and before general anesthesia wears off,
  Interventions: Device: Immediate urinary catheter removal
- UC removal within 24hr after surgery (Active Comparator): A urinary catheter is removed in the ward within postoperative 1 day (within 24 hours after surgery).
  Interventions: Device: urinary catheter removal within postoperative 1day

INTERVENTIONS:
Device: Immediate urinary catheter removal — A urinary catheter is removed immediately after surgery and before general anesthesia wears off in the operating room.
  Arms: Immediate UC removal after surgery
Device: urinary catheter removal within postoperative 1day — The urethral catheter will be removed in the ward within 1 day after surgery (within 24 hours after surgery).
  Arms: UC removal within 24hr after surgery

SUMMARY:
The enhanced recovery after surgery (ERAS) program is widely applied in colorectal cancer surgery. Among the early recovery programs after surgery, the timing of removal of the urinary catheter after surgery has been emphasized recently, but the specific timing is still under discussion. Maintaining the urinary catheter after surgery is to prevent urinary retention after surgery, but it is known that the risk of urinary tract infection increases the longer it is maintained. Previously, it was removed 3 days after colorectal cancer surgery, but several studies reported that even if it was removed earlier, the incidence of urinary retention did not increase, and rather the incidence of urinary tract infection decreased. In particular, by applying the early recovery program after surgery, factors related to patient recovery before, during, and after surgery are applied to help rapid recovery, and it has been reported that early removal of the urinary catheter has a positive effect on postoperative recovery and complications. Therefore, it is necessary to prove that the timing of removal of the urinary catheter after surgery in colorectal cancer patients can help early recovery through clinical results such as patient recovery and occurrence of complications.

DETAILED DESCRIPTION:
This study aims to demonstrate that removing the urinary drain immediately after colorectal cancer surgery is non-inferior to removing it on the first day (within 24 hours) after surgery in terms of the incidence of acute urinary retention.

To evaluate the non-inferiority of the incidence of acute urinary retention (AUR) according to the timing of urinary drain removal after surgery.

Secondary outcomes are the incidence of symptomatic urinary tract infection (UTI), postvoid residual (PVR), length of hospital stay, postoperative pain score, and narcotic analgesic usage, early ambulation success rate, postoperative complication rate, and overactive bladder symptom assessment score for patient discomfort, etc., and to compare the clinical outcomes after surgery from various perspectives.

ELIGIBILITY:
Inclusion Criteria:

* 19 years old 80 years old
* Patients diagnosed with colorectal cancer who are eligible for radical resection surgery
* Patients who underwent open, laparoscopic, or robotic surgery
* Written informed consent

Exclusion Criteria:

* Patients who have undergone two or more major abdominal surgeries, including lateral pelvic lymph node dissection, at the same time
* Patients who require continuous monitoring through a urinary catheter due to hemodynamic instability or massive bleeding, etc.
* Patients who have undergone conventional treatment in cases other than distant metastasis or R0 resection
* Patients who have developed complications related to the urinary system during surgery and require maintenance of a urinary catheter such as a urethral stent
* Patients who have undergone urinary surgery such as urethral stent placement, cystectomy, or urostomy in the past
* Patients who are on hemodialysis or peritoneal dialysis due to chronic renal failure
* Patients who cannot participate in a clinical trial at the discretion of a physician
* Patients who do not wish to participate in the study

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute urinary retention due to failure to void spontaneously within 4 hours after removal of a urinary drain | 3 days after surgery
  - Definition of acute urinary retention: Failure to urinate spontaneously within 4 hours after removal of the urinary drainage tube or occurrence of residual volume greater than 400 ml as measured by ultrasound

SECONDARY OUTCOMES:
Incidence of urinary drainage tube reinsertion rates | 7 days after surgery
  The rate of re-insertion of a urinary catheter due to failure of self-voiding at 4 hours after surgery and re-evaluation 4 hours later according to the protocol
Incidence of symptomatic urinary tract infections (UTIs) | 30 days postoperatively
  Bacterial identification rate of 10^5 CFU/mL or higher in urine culture test with clinical symptoms
postoperative pain scores | 3 days after surgery
  Visual analog scale (VAS) score at 4±2 hours, 24±6 hours, and 48±6 hours after surgery.
  The NRS is a single-item scale in which patients choose a number from 0 to 10 that best represents their pain intensity, with 0 indicating no pain, 1 to 3 indicating mild pain, 4 to 6 indicating moderate pain, and 7 to 10 indicating severe pain .
Postoperative narcotic analgesic use rate | 3 days after surgery
  Rates of narcotic analgesic use at 4±2 hours, 24±6 hours, and 48±6 hours postoperatively
early walking success rates | 3 days after surgery
  Success rate of walking for more than 15 minutes three times a day at 4±2 hours, 24±6 hours, and 48±6 hours after surgery
postoperative complications | 30 days after surgery
  Charlson comorbidity index (CCI) score within 1 month of discharge from surgery. The CCI is based on the Clavien system but accounts for all accumulated complications and provides a continuous overall score between 0-100. The higher the score, the worse it is.
Evaluation of patient symptom and quality of life | 30 days after surgery
  Comparison of overactive bladder symptom assessment scores. Patient evaluation is performed using the Overactive Bladder Questionnaire (OAB-q short form) questionnaire. It consists of 19 items, each item is evaluated from 1 to 6 points, and the total score is 114 points. A higher score indicates more discomfort from overactive bladder.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St.Mary's hospital, the Catholic university of Korea, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No